CLINICAL TRIAL: NCT05770453
Title: Evaluation of the Presence of a Double Anaerobic Threshold in a Population of Athletes
Brief Title: Double Anaerobic Threshold in Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other); University of Foggia (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1719
Record Dates: First submitted 2023-02-21; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Cardiopulmonary Exercise Test; Anaerobic Threshold; Athlete

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During an incremental cardiopulmonary exercise test (CPET) performed with a ramp protocol, it is very important to determine the anaerobic threshold, defined as the point at which the metabolism switches from being predominantly aerobic to also being anaerobic. The anaerobic threshold can be determined invasively, by identifying the increase in blood lactates with an arterial sampling, or, more commonly, non-invasively by three methods: the V-slope method, the ventilatory equivalents method and by using end-expiratory oxygen and carbon dioxide pressure (PETO2 and PETCO2 respectively). Normally, the anaerobic threshold is determined by the first method and the other two are used to confirm the value. The finding of different anaerobic threshold values using these three methods has been reported anecdotally in the past, while a prevalence of 11% in a healthy population has recently been described. Regular training, particularly that aimed at endurance sports, is able to shift the anaerobic threshold to higher exercise intensities. At present, the physiological reasons for the presence of a double threshold are unclear.

The aim of the study is to identify the anaerobic threshold by means of the V-slope method and by means of the ventilatory equivalents method in athletes who have performed an incremental ramp CPET at the laboratories of the investigating centres, to assess in how many athletes a double threshold is present and to try to interpret the physiological/ pathophysiological significance of this finding.

In this retrospective and prospective observational study, healthy male and female athletes who have had a cardiopulmonary test at our laboratories from 2007 to the present (retrospectively recruited) and prospectively recruited until the calculated sample size is reached will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* no major present or past illnesses, no ongoing treatment
* At least 2 training sessions per week.

Exclusion Criteria:

* Current illnesses and treatments for any physical condition that could potentially alter performance
* Subjects who have performed a submaximal test (RER < 1.05)
* CPET during which the AT determination is poorly assessable, i.e. due to changes in respiration.
* obese subjects (BMI >30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female athletes who performed a cardiopulmonary test at our laboratories from 2007 to the present (retrospectively recruited) and prospectively recruited will be enrolled
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Athletes groups | immediately after the incremental cardiopulmonary exercise test evaluation
  Identification of two groups of athletes (those with identified double anaerobic threshold and those without)

SECONDARY OUTCOMES:
Groups differences in age | immediately after the incremental cardiopulmonary exercise test evaluation
  Assess whether there are differences in age (years) between the two groups of subjects.
Groups differences in sport practised | immediately after the incremental cardiopulmonary exercise test evaluation
  Assess whether the two groups of subjects differ in term of the sport practised (information collected during patient interview)
Groups differences in exercise performance | immediately after the incremental cardiopulmonary exercise test evaluation
  Assess whether the two groups of subjects differ in term of exercise performance (peak power (Watts) reached during CPET)
Groups differences in VO2 | immediately after the incremental cardiopulmonary exercise test evaluation
  Assess whether there are differences in the oxygen intake VO2 (cardiopulmonary exercise test) between the two groups
Groups differences in VE/VCO2 slope | immediately after the incremental cardiopulmonary exercise test evaluation
  Assess whether there are differences in minute ventilation/carbon dioxide production relationship VE/VCO2 slope (cardiopulmonary exercise test) between the two groups
Groups differences in VE | immediately after the incremental cardiopulmonary exercise test evaluation
  Assess whether there are differences in minute ventilation VE (cardiopulmonary exercise test) between the two groups
Differences in VO2 at the two thresholds | immediately after the incremental cardiopulmonary exercise test evaluation
  Highlight the differences in oxygen intake VO2 (cardiopulmonary exercise test), in the subjects with double anaerobic threshold, at the two thresholds.
Differences in VE/VCO2 at the two thresholds | immediately after the incremental cardiopulmonary exercise test evaluation
  Highlight the differences in minute ventilation/carbon dioxide production relationship VE/VCO2 slope (cardiopulmonary exercise test), in the subjects with double anaerobic threshold, at the two thresholds.
Differences in VE at the two thresholds | immediately after the incremental cardiopulmonary exercise test evaluation
  Highlight the differences in minute ventilation VE (cardiopulmonary exercise test), in the subjects with double anaerobic threshold, at the two thresholds.

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, Prof., Principal Investigator — Centro Cardiologico Monzino
Locations (3):
- Italy (3):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - University of Foggia, Foggia
  - Centro Cardiologico Monzino, Milan

IPD SHARING:
Plan to Share IPD: Undecided